CLINICAL TRIAL: NCT03645421
Title: A Phase IIa, Randomised, Parallel, Double-Blind,Placebo-Controlled Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of MEDI0382 in Japanese Preobese or Obese Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: Safety and Tolerability Study of MEDI0382 in Japanese Preobese or Obese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5674C00001
Record Dates: First submitted 2018-06-25; First posted 2018-08-24 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; MEDI0382; D5674C00001; T2DM; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo (Placebo Comparator): Placebo per day,SC injection on 48 days.
  Interventions: Drug: PlaceboA; Drug: PlaceboB
- MEDI0382 100μg (Experimental): 50 μg/day,SC injection on the first 5 days and 100 μg/day,SC injection on 43 days
  Interventions: Drug: MEDI0382 100 μg; Drug: MEDI0382 50 ug
- MEDI0382 200μg (Experimental): 50 μg/day,SC injection on the first 5 days, 100 μg/day,SC injection on 7 days and 200 μg/day,SC injection on 36 days.
  Interventions: Drug: MEDI0382 100 μg; Drug: MEDI0382 200 μg; Drug: MEDI0382 50 ug
- MEDI0382 300μg (Experimental): 50 μg/day,SC injection on the first 5 days, 100 μg/day,SC injection on 7 days, 200 μg/day,SC injection on 7 days and 300 μg/day,SC injection on 29 days
  Interventions: Drug: MEDI0382 100 μg; Drug: MEDI0382 200 μg; Drug: MEDI0382 300 μg; Drug: MEDI0382 50 ug

INTERVENTIONS:
Drug: MEDI0382 100 μg — Solution for injection in 1.0 mL pre-filled syringe, 100 μg per dose, 1 dose
  Arms: MEDI0382 100μg; MEDI0382 200μg; MEDI0382 300μg
Drug: MEDI0382 200 μg — Solution for injection in 1.0 mL pre filled syringe 200 μg per dose, 1 dose
  Arms: MEDI0382 200μg; MEDI0382 300μg
Drug: MEDI0382 300 μg — Solution for injection in 1.0 mL pre filled syringe, 300 μg per dose, 1 dose
  Arms: MEDI0382 300μg
Drug: PlaceboA — 1.0 mL liquid formulation per Vial
  Arms: placebo
Drug: MEDI0382 50 ug — Solution for injection, 1.0 mL per vial, 50 ug
  Arms: MEDI0382 100μg; MEDI0382 200μg; MEDI0382 300μg
Drug: PlaceboB — Solution for injection in 1.0 mL pre-filled syringe.
  Arms: placebo

SUMMARY:
This is a Phase 2a study designed to assess the safety and tolerability of MEDI0382 titrated up to a dose level of 100, 200 or 300 µg from 50 µg vs Placebo across 48 days in Japanese subjects.

The study D5674C00001 can be conducted with a reasonable expectation of safety and tolerability in Japanese T2DM patients. The design of this study has taken into account the known benefits and risks of GLP-1 receptor agonists and glucagon receptor agonists as well as the translatable effects observed in nonclinical studies of MEDI0382.

DETAILED DESCRIPTION:
This is a randomized, parallel-group, placebo-controlled, double-blind, multicenter Phase Ⅱa study to evaluate the safety, efficacy, and pharmacokinetics of MEDI0382 in Japanese preobese and obese subjects with type 2 diabetes who have inadequate glycemic control with diet and exercise. Subject fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomised in a 1:1:1:1 ratio to four treatment arms. This is a Phase IIa study designed to evaluate the dose range for MEDI0382 to explore the safety profile, as well as blood glucose control and weight loss effects of MEDI0382 in Japanese patients with T2DM. The design of this study has taken into account the known benefits and risks of GLP-1 receptor agonists and glucagon receptor agonists as well as the translatable effects observed in nonclinical studies of MEDI0382, such that benefit-risk balance for the Japanese preobese and obese patients with T2DM in this study is considered favourable. A treatment period of 48 days is required to properly evaluate the dose range and safety and tolerability in three different doses. Inclusion of placebo in the study allows appropriate basis of AEs, glycaemic control, and weight loss. Benefits related to participation in this trial include close follow-up of a subject's diabetes and treatment with anti-diabetes agents. Although one of possible treatments is placebo, appropriate rescue therapy for worsening glycaemic control will be implemented if required.

ELIGIBILITY:
Inclusion Criteria:

* Individuals whose HbA1c range of 7.0% to 10.5% (inclusive) at screening.
* Individuals who are diagnosed with T2DM
* Individuals whose current condition at enrolment (Visit 1) is drug naïve
* BMI within the range of 24 - 40 kg/m2 (inclusive) at screening

Exclusion Criteria:

* Subjects with any of the following results at screening:
* Aspartate transaminase (AST) ≥ 2.5 × upper limit of normal (ULN)
* Alanine transaminase (ALT) ≥ 2.5 × ULN
* Total bilirubin (TBL) ≥ 2 × ULN
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) ≤ 60 mL/minute/1.73 m2 at screening
* Participation in another clinical study with an investigational product administered in the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi

REFERENCES:
- See also: d5674c00001 CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5674C00001&attachmentIdentifier=178319f5-5ef4-4cca-856f-fdfb344927ae&fileName=d5674c00001_CSP_redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5674C00001&attachmentIdentifier=725e1184-cf38-400c-bd99-3105851a5afa&fileName=d5674c00001_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Preobese/obese Japanese adults with Type 2 diabetes mellitus (T2DM) were recruited to this Phase IIa randomised, parallel-group, placebo-controlled, double-blind, study at 5 centres in Japan. The first patient started in August 2018 and the last patient completed in January 2019.
Pre-assignment Details: Patients with an early stage of T2DM who had inadequate blood glucose control, defined as glycated haemoglobin (HbA1c) between 7.0% and 10.5%, and who were treated with diet and exercise were enrolled. A body mass index of 24 to 40 kg/m2 was also a requirement. Patients with acutely decompensated blood glucose control were excluded.
Groups:
- Placebo: Patients were randomised to receive MEDI0382 matched placebo for 48 days.
- MEDI0382 100 mcg: Patients were randomised to receive 100 micrograms (mcg) MEDI0382 per day by subcutaneous (SC) injection, titrated as follows: 50 mcg/day for 5 days and then 100 mcg/day for 43 days.
- MEDI0382 200 mcg: Patients were randomised to receive 200 mcg MEDI0382 per day by SC injection, titrated as follows: 50 mcg/day for 5 days, 100 mcg/day for 7 days and then 200 mcg/day for 36 days.
- MEDI0382 300 mcg: Patients were randomised to receive 300 mcg MEDI0382 per day by SC injection, titrated as follows: 50 mcg/day for 5 days, 100 mcg/day for 7 days, 200 mcg/day for 7 days and then 300 mcg/day for 29 days.
Period: Overall Study
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Started | 16 | 15 | 15 | 15
Received Investigational Product (IP) | 16 | 15 | 15 | 15
Completed | 16 | 15 | 10 | 11
Not Completed | 0 | 0 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 4 | 1
Not completed — Withdrawal by patient | 0 | 0 | 0 | 3
Not completed — Study specific withdrawal criteria | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the Full Analysis Set which included all randomised patients who received at least 1 dose of IP, analysed according to their randomised treatment group.
Groups:
- MEDI0382 100 mcg: Patients were randomised to receive 100 mcg MEDI0382 per day by SC injection, titrated as follows: 50 mcg/day for 5 days and then 100 mcg/day for 43 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg | Total
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (8.6) | 56.7 (10.7) | 58.7 (11.3) | 57.5 (9.2) | 58.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 2 | 2 | 14
  Male | 13 | 8 | 13 | 13 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 16 | 15 | 15 | 15 | 61
  Not Hispanic or Latino | 16 | 15 | 15 | 15 | 61

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in 24-Hour Heart Rate at Days 20 and 48
Description: Twenty four-hour heart rate was determined using an ambulatory blood pressure monitoring (ABPM) device, and the mean change from baseline in the 24-hour heart rate is presented for Days 20 and 48.
Time Frame: Baseline (Day -1) and Days 20 and 48.
Population: The Safety Analysis Set included all randomised patients who received at least 1 dose of IP, analysed according to the treatment received. Patients with data available at each timepoint are presented.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
beats/minute
  Day 20: number analyzed (Participants) | 15 | 15 | 12 | 12
  Day 20 | -1.86 (7.43) | 6.65 (7.46) | 13.50 (5.86) | 15.80 (7.86)
  Day 48: number analyzed (Participants) | 15 | 15 | 8 | 9
  Day 48 | -0.25 (7.24) | 7.87 (8.60) | 12.81 (4.93) | 15.22 (5.50)

2. Primary Outcome: Mean Change From Baseline in 24-Hour Systolic and Diastolic Blood Pressure (BP) at Days 20 and 48
Description: Twenty four-hour BP was determined using an ABPM device, and the mean change from baseline in the 24-hour systolic BP and 24-hour diastolic BP are presented for Days 20 and 48.
Time Frame: Baseline (Day -1) and Days 20 and 48.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimetres of mercury
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
millimetres of mercury
  24-hour Systolic BP: Day 20: number analyzed (Participants) | 15 | 15 | 12 | 12
  24-hour Systolic BP: Day 20 | 2.98 (9.00) | -4.09 (8.93) | -7.24 (10.54) | -2.48 (9.28)
  24-hour Systolic BP: Day 48: number analyzed (Participants) | 15 | 15 | 8 | 9
  24-hour Systolic BP: Day 48 | 0.08 (14.32) | -2.27 (12.42) | -5.17 (19.35) | -6.97 (7.48)
  24-hour Diastolic BP: Day 20: number analyzed (Participants) | 15 | 15 | 12 | 12
  24-hour Diastolic BP: Day 20 | 0.98 (4.34) | -0.62 (3.42) | -1.41 (4.56) | 0.81 (5.58)
  24-hour Diastolic BP: Day 48: number analyzed (Participants) | 15 | 15 | 8 | 9
  24-hour Diastolic BP: Day 48 | -0.06 (6.82) | -0.66 (4.56) | -0.27 (9.17) | -0.68 (3.88)

3. Primary Outcome: Mean Percentage Change From Baseline in Glucose Area Under the Plasma Concentration Curve (AUC[0-4h]) as Measured by a Standardised Mixed-Meal Test (MMT) at Day 48
Description: The MMT was conducted following a minimum 8-hour fast. Blood samples for glucose monitoring were taken 15 minutes before the patient consumed a standardised meal, and samples were taken at intervals after the meal, up to 4 hours. The MMT glucose AUC(0-4h) was calculated using a trapezoidal method, and the mean percentage change from baseline at Day 48 was analysed using an analysis of covariance (ANCOVA) model with treatment group as a factor and baseline as a covariate.
Time Frame: Baseline (Day -1) and Day 48: 15 minutes before standardised meal, and then at 15, 30, 45, 60, 90, 120, 180 and 240 minutes (+/-5 minutes) after consumption of the standardised meal.
Population: The Full Analysis Set included all randomised patients who received at least 1 dose of IP, analysed according to their randomised treatment group. MMTs were not conducted on patients who prematurely discontinued IP.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Percentage change | 2.45 [-3.37 to 8.26] | -39.66 [-45.67 to -33.66] | -31.16 [-38.61 to -23.71] | -37.86 [-44.95 to -30.76]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Pair-wise comparison of MEDI0382 100 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; Least squares (LS) mean difference = -42.11, 95% CI 2-sided [-50.47 to -33.75], Standard Error of Mean 4.16 — Treatment difference = MEDI0382 100 mcg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Pair-wise comparison of MEDI0382 200 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -33.61, 95% CI 2-sided [-43.04 to -24.18], Standard Error of Mean 4.69 — Treatment difference = MEDI0382 200 mcg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Pair-wise comparison of MEDI0382 300 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -40.30, 95% CI 2-sided [-49.49 to -31.12], Standard Error of Mean 4.57 — Treatment difference = MEDI0382 300 mcg - Placebo

4. Primary Outcome: Mean Percentage Change From Baseline in Body Weight at Day 48
Description: The mean percentage change from baseline in body weight at Day 48 was analysed using an ANCOVA model with treatment group as a factor and baseline as a covariate. For patients who prematurely discontinued IP, the last on-treatment measurement, regardless of rescue medication, was used (last observation carried forward [LOCF]).
Time Frame: Baseline (Day -1) and Day 48.
Population: The Full Analysis Set included all randomised patients who received at least 1 dose of IP, analysed according to their randomised treatment group. Patients with data available are presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Percentage change | -0.82 [-2.06 to 0.43] | -2.12 [-3.40 to -0.84] | -3.34 [-4.68 to -2.01] | -3.34 [-4.61 to -2.06]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Pair-wise comparison of MEDI0382 100 mcg versus Placebo; Test type: Other; p = 0.1476, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -1.30, 95% CI 2-sided [-3.08 to 0.47], Standard Error of Mean 0.89 — Treatment difference = MEDI0382 100 mcg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Pair-wise comparison of MEDI0382 200 mcg versus Placebo; Test type: Other; p = 0.0080, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -2.53, 95% CI 2-sided [-4.37 to -0.69], Standard Error of Mean 0.92 — Treatment difference = MEDI0382 200 mcg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Pair-wise comparison of MEDI0382 300 mcg versus Placebo; Test type: Other; p = 0.0063, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -2.52, 95% CI 2-sided [-4.30 to -0.74], Standard Error of Mean 0.89 — Treatment difference = MEDI0382 300 mcg - Placebo

5. Primary Outcome: Mean Change From Baseline in Heart Rate Measured by Electrocardiogram (ECG) at Day 48.
Description: Digital ECGs were taken at baseline and predose and postdose on Days 1, 6, 13, 20 and 48. The mean change from baseline is presented.
Time Frame: Baseline (Day -1) and Days 1, 6, 13, 20 and 48: predose and 6 hours (+/-15 minutes) postdose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
beats/minute
  Day 1: 6 hours postdose | 1.77 (7.20) | 4.24 (5.00) | 2.18 (8.62) | 6.27 (7.91)
  Day 6: predose: number analyzed (Participants) | 16 | 15 | 14 | 14
  Day 6: predose | -2.85 (4.93) | 1.84 (8.56) | 7.69 (7.11) | 10.79 (5.87)
  Day 6: 6 hours postdose: number analyzed (Participants) | 16 | 15 | 14 | 14
  Day 6: 6 hours postdose | 0.02 (8.79) | 4.62 (9.11) | 8.88 (6.06) | 10.67 (7.59)
  Day 13: predose: number analyzed (Participants) | 16 | 15 | 14 | 13
  Day 13: predose | -2.63 (5.58) | 6.91 (8.83) | 8.93 (6.84) | 11.74 (7.92)
  Day 13: 6 hours postdose: number analyzed (Participants) | 16 | 15 | 14 | 13
  Day 13: 6 hours postdose | 2.19 (9.13) | 6.40 (11.41) | 16.62 (7.14) | 13.31 (9.45)
  Day 20: predose: number analyzed (Participants) | 16 | 15 | 13 | 12
  Day 20: predose | -1.85 (7.52) | 6.24 (8.02) | 11.97 (8.12) | 13.03 (8.65)
  Day 20: 6 hours postdose: number analyzed (Participants) | 16 | 15 | 13 | 12
  Day 20: 6 hours postdose | 0.29 (9.15) | 5.09 (9.37) | 16.79 (6.21) | 16.94 (8.86)
  Day 48: predose: number analyzed (Participants) | 16 | 15 | 10 | 11
  Day 48: predose | -1.06 (10.06) | 7.20 (5.88) | 10.20 (9.70) | 17.06 (6.12)
  Day 48: 6 hours postdose: number analyzed (Participants) | 16 | 15 | 10 | 11
  Day 48: 6 hours postdose | -6.25 (10.34) | 1.16 (10.21) | 15.43 (12.15) | 12.70 (5.95)

6. Primary Outcome: Number of Patients Who Experienced Adverse Events (AEs)
Description: AEs were collected from Day 1 of treatment up to 14 days after the last dose of IP. Serious AEs (SAEs) were collected from signing of informed consent. The numbers of patients who experienced any AE, any SAE (including events with an outcome of death), and any AE leading to discontinuation of IP are presented.
Time Frame: Day 1 up to 14 days after the last dose of IP (approximately 9 weeks).
Population: The Safety Analysis Set included all randomised patients who received at least 1 dose of IP, analysed according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Participants
  Any AE | 6 | 6 | 11 | 9
  Any SAE | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of IP | 0 | 0 | 4 | 1

7. Secondary Outcome: Mean Change From Baseline in HbA1c at Day 48
Description: The mean change from baseline in HbA1c at Day 48 was analysed using an ANCOVA model with treatment group as a factor and baseline as a covariate. For patients who prematurely discontinued IP, or for patients who did not have a measurement taken on Day 48, the last post-baseline measurement, regardless of rescue medication, was used (LOCF).
Time Frame: Baseline (Day -1) and Day 48 (predose).
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent glycated haemoglobin
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Percent glycated haemoglobin | -0.14 [-0.41 to 0.12] | -1.23 [-1.51 to -0.96] | -1.24 [-1.53 to -0.96] | -0.90 [-1.18 to -0.63]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Pair-wise comparison of MEDI0382 100 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -1.09, 95% CI 2-sided [-1.48 to -0.70], Standard Error of Mean 0.19 — Treatment difference = MEDI0382 100 mcg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Pair-wise comparison of MEDI0382 200 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -1.10, 95% CI 2-sided [-1.49 to -0.71], Standard Error of Mean 0.19 — Treatment difference = MEDI0382 200 mcg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Pair-wise comparison of MEDI0382 300 mcg versus Placebo; Test type: Other; p = 0.0002, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -0.76, 95% CI 2-sided [-1.15 to -0.38], Standard Error of Mean 0.19 — Treatment difference = MEDI0382 300 mcg - Placebo

8. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose at Day 48
Description: The mean change from baseline in fasting plasma glucose at Day 48 was analysed using an ANCOVA model with treatment group as a factor and baseline as a covariate. For patients who prematurely discontinued IP, or for patients who did not have a measurement taken on Day 48, the last post-baseline measurement, regardless of rescue medication, was used (LOCF).
Time Frame: Baseline (Day -1) and Day 48 (predose).
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per decilitre (mg/dL)
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
milligrams per decilitre (mg/dL) | -0.40 [-12.60 to 11.80] | -57.10 [-69.77 to -44.42] | -60.98 [-76.82 to -45.15] | -55.47 [-70.28 to -40.66]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Pair-wise comparison of MEDI0382 100 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -56.69, 95% CI 2-sided [-74.30 to -39.09], Standard Error of Mean 8.75 — Treatment difference = MEDI0382 100 mcg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Pair-wise comparison of MEDI0382 200 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -60.58, 95% CI 2-sided [-80.53 to -40.63], Standard Error of Mean 9.92 — Treatment difference = MEDI0382 200 mcg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Pair-wise comparison of MEDI0382 300 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -55.07, 95% CI 2-sided [-74.28 to -35.86], Standard Error of Mean 9.55 — Treatment difference = MEDI0382 300 mcg - Placebo

9. Secondary Outcome: Mean Change From Baseline in Fructosamine at Day 48
Description: The mean change from baseline in fructosamine at Day 48 was analysed using an ANCOVA model with treatment group as a factor and baseline as a covariate. For patients who prematurely discontinued IP, the last on-treatment measurement, regardless of rescue medication, was used (LOCF).
Time Frame: Baseline (Day -1) and Day 48 (predose).
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per litre (mmol/L)
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
millimoles per litre (mmol/L) | -0.012 [-0.029 to 0.004] | -0.083 [-0.100 to -0.066] | -0.066 [-0.083 to -0.048] | -0.061 [-0.079 to -0.044]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Pair-wise comparison of MEDI0382 100 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -0.071, 95% CI 2-sided [-0.094 to -0.047], Standard Error of Mean 0.012 — Treatment difference = MEDI0382 100 mcg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Pair-wise comparison of MEDI0382 200 mcg versus Placebo; Test type: Other; p < 0.0001, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -0.053, 95% CI 2-sided [-0.077 to -0.030], Standard Error of Mean 0.012 — Treatment difference = MEDI0382 200 mcg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Pair-wise comparison of MEDI0382 300 mcg versus Placebo; Test type: Other; p = 0.0002, ANCOVA; Analysis used treatment group as a factor and baseline as a covariate; LS mean difference = -0.049, 95% CI 2-sided [-0.074 to -0.024], Standard Error of Mean 0.012 — Treatment difference = MEDI0382 300 mcg - Placebo

10. Secondary Outcome: Mean Change From Baseline in the Percentage of Time in Hyperglycaemia Over 24 Hours at Days 5, 12, 19 and 47
Description: Hyperglycaemia was defined as blood glucose >7.8 mmol/L or >140 mg/dL. Continuous glucose monitoring used a device fitted to the upper arm by trained study site staff to measure and record interstitial glucose levels every 15 minutes. Analysis was based on 24-hour readings defined as the first available time point with a valid continuous glucose monitoring glucose reading. The change in the percentage time in hyperglycaemia from the last day of baseline continuous glucose monitoring over 24 hours to the end of dosing at each dose level for the indicated timepoints is presented.
Time Frame: Baseline (Day -8 to -2) and Days 5, 12, 19 and 47.
Population: The Full Analysis Set included all randomised patients who received at least 1 dose of IP, analysed according to their randomised treatment group. Patients with data available at each time point are presented.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Percentage of time
  Day 5: number analyzed (Participants) | 13 | 15 | 13 | 7
  Day 5 | -3.23 (12.59) | -48.35 (21.27) | -33.71 (24.67) | -51.33 (30.04)
  Day 12: number analyzed (Participants) | 12 | 14 | 10 | 8
  Day 12 | -11.72 (28.58) | -57.74 (24.59) | -53.36 (21.59) | -55.78 (25.19)
  Day 19: number analyzed (Participants) | 10 | 14 | 12 | 9
  Day 19 | -12.08 (17.61) | -59.57 (16.98) | -43.85 (28.96) | -60.68 (24.93)
  Day 47: number analyzed (Participants) | 11 | 15 | 9 | 6
  Day 47 | -6.15 (22.80) | -47.99 (20.63) | -48.96 (20.28) | -57.59 (21.86)

11. Secondary Outcome: Mean Change From Baseline in the Percentage of Time in Hypoglycaemia Over 24 Hours at Days 5, 12, 19 and 47
Description: Hypoglycaemia was defined as blood glucose <3 mmol/L or <54 mg/dL. Continuous glucose monitoring used a device fitted to the upper arm by trained study site staff to measure and record interstitial glucose levels every 15 minutes. Analysis was based on 24-hour readings defined as the first available time point with a valid continuous glucose monitoring glucose reading. The change in the percentage time in hypoglycaemia from the last day of baseline continuous glucose monitoring over 24 hours to the end of dosing at each dose level for the timepoints is presented.
Time Frame: Baseline (Day -8 to -2) and Days 5, 12, 19 and 47.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Percentage of time
  Day 5: number analyzed (Participants) | 13 | 15 | 13 | 7
  Day 5 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 6.28 (16.61)
  Day 12: number analyzed (Participants) | 12 | 14 | 10 | 8
  Day 12 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 19: number analyzed (Participants) | 10 | 14 | 12 | 9
  Day 19 | 0.00 (0.00) | 0.00 (0.00) | 3.68 (12.75) | 0.00 (0.00)
  Day 47: number analyzed (Participants) | 11 | 15 | 9 | 6
  Day 47 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

12. Secondary Outcome: Mean Change From Baseline in the Percentage of Time in Hyperglycaemia Over 5 Days for 50 mcg Dose Level and 7 Days for Other Dose Levels
Description: Hyperglycaemia was defined as blood glucose >7.8 mmol/L or >140 mg/dL. Continuous glucose monitoring used a device fitted to the upper arm by trained study site staff to measure and record interstitial glucose levels every 15 minutes. Analysis was based on 24-hour readings defined as the first available time point with a valid continuous glucose monitoring glucose reading. The change in the percentage time in hyperglycaemia from the last day of baseline continuous glucose monitoring over 5 days for 50 mcg MEDI0382 and 7 days for each of the dose levels (during titration) is presented, up to Day 47, per randomised group.
Time Frame: Baseline (Day -8 to -2) and Days 1 to 5, 6 to 12, 13 to 19 and 41 to 47.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Percentage of time
  Days 1 to 5: number analyzed (Participants) | 13 | 14 | 12 | 9
  Days 1 to 5 | -1.43 (10.26) | -42.52 (13.46) | -38.68 (18.97) | -34.74 (18.24)
  Days 6 to 12: number analyzed (Participants) | 12 | 15 | 10 | 9
  Days 6 to 12 | -8.97 (26.12) | -48.35 (16.01) | -50.81 (18.97) | -51.82 (16.73)
  Days 13 to 19: number analyzed (Participants) | 12 | 15 | 12 | 10
  Days 13 to 19 | -6.09 (19.10) | -53.25 (16.47) | -52.33 (20.96) | -47.50 (20.67)
  Days 41 to 47: number analyzed (Participants) | 11 | 15 | 10 | 8
  Days 41 to 47 | -0.40 (22.70) | -42.37 (17.22) | -43.44 (18.26) | -51.25 (17.12)

13. Secondary Outcome: Mean Change From Baseline in the Percentage of Time in Hypoglycaemia Over 5 Days for 50 mcg Dose Level and 7 Days for Other Dose Levels
Description: Hyp0glycaemia was defined as blood glucose <3 mmol/L or <54 mg/dL. Continuous glucose monitoring used a device fitted to the upper arm by trained study site staff to measure and record interstitial glucose levels every 15 minutes. Analysis was based on 24-hour readings defined as the first available time point with a valid continuous glucose monitoring glucose reading. The change in the percentage time in hypoglycaemia from the last day of baseline continuous glucose monitoring over 5 days for 50 mcg MEDI0382 and 7 days for each of the randomised dose levels (during titration) is presented, up to Day 47, per randomised group.
Time Frame: Baseline (Day -8 to -2) and Days 1 to 5, 6 to 12, 13 to 19 and 41 to 47.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 16 | 15 | 15 | 15
Percentage of time
  Days 1 to 5: number analyzed (Participants) | 13 | 14 | 12 | 9
  Days 1 to 5 | 0.21 (0.76) | 0.06 (0.27) | 0.25 (0.55) | 5.50 (16.57)
  Days 6 to 12: number analyzed (Participants) | 12 | 15 | 10 | 9
  Days 6 to 12 | 0.06 (0.22) | 0.90 (2.24) | 0.07 (0.19) | 0.13 (0.62)
  Days 13 to 19: number analyzed (Participants) | 12 | 15 | 12 | 10
  Days 13 to 19 | 0.10 (0.30) | 0.41 (1.25) | 2.97 (5.43) | 1.09 (1.58)
  Days 41 to 47: number analyzed (Participants) | 11 | 15 | 10 | 8
  Days 41 to 47 | 0.01 (0.04) | -0.02 (0.05) | 0.30 (0.60) | 2.59 (7.22)

14. Secondary Outcome: Mean Trough Plasma Concentration (Ctrough) of MEDI0382 up to Day 48
Description: To evaluate pharmacokinetics (PK), blood samples were collected predose and Ctrough of MEDI0382 was determined. Results are presented for Days 2, 5, 34 and 48.
Time Frame: Blood samples collected predose on Days 1 to 6, 13, 20, 34 and 48.
Population: The PK Analysis Set included all patients who received at least 1 dose of MEDI0382 and had at least 1 post-baseline MEDI0382 PK sample taken that was above the lower limit of quantification. Patients with data available at each timepoint are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre
Arm/Group | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 15 | 15 | 15
nanograms per millilitre
  Day 2 | 1.20 (41.8) | 1.22 (22.9) | 1.11 (26.9)
  Day 5: number analyzed (Participants) | 15 | 14 | 14
  Day 5 | 1.47 (36.8) | 1.61 (26.6) | 1.56 (25.8)
  Day 34: number analyzed (Participants) | 15 | 11 | 11
  Day 34 | 2.70 (78.0) | 5.16 (81.4) | 7.18 (39.8)
  Day 48: number analyzed (Participants) | 15 | 10 | 11
  Day 48 | 2.83 (77.5) | 7.14 (23.8) | 9.12 (24.7)

15. Secondary Outcome: Number of Patients With Antidrug Antibody (ADA) Response to MEDI0382
Description: The number of patients who were ADA positive at baseline and/or post-baseline are presented. Persistent positive was defined as positive at ≥2 post-baseline assessments (with ≥16 weeks between first and last positive) or positive at the last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive.
  +ve = positive
Time Frame: Samples were collected predose on days 1, 13, 20 and 48, and 7 to 14 days after administration of last dose of IP.
Population: The PK Analysis Set included all patients who received at least 1 dose of MEDI0382 and had at least 1 post-baseline MEDI0382 PK sample taken that was above the lower limit of quantification.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 15 | 15 | 15
Participants
  ADA +ve at baseline | 0 | 0 | 0
  ADA +ve post-baseline | 4 | 5 | 2
  ADA +ve post-baseline & +ve at baseline | 0 | 0 | 0
  ADA+ve post-baseline & not detected at baseline | 4 | 5 | 2
  Persistent +ve | 2 | 4 | 2
  Transient +ve | 2 | 1 | 0
  ADA not detected post-baseline & +ve baseline | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected from Day 1 of treatment up to 14 days after the last dose of IP (approximately 9 weeks).
Description: AEs are presented for the Safety Analysis Set which included all randomised patients who received at least 1 dose of IP, analysed according to the treatment received.
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 6/16 | 6/15 | 11/15 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | MEDI0382 100 mcg (N=15) | MEDI0382 200 mcg (N=15) | MEDI0382 300 mcg (N=15)
Nausea (Gastrointestinal disorders) | 1 | 2 | 7 | 4
Vomiting (Gastrointestinal disorders) | 0 | 3 | 5 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 3
Injection site bruising (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI needs to provide sponsor with the draft to review no later than 30 days prior to the date of publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03645421/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03645421/SAP_001.pdf